CLINICAL TRIAL: NCT06271408
Title: Xenon Xe 129 Hyperpolarized MRI Ventilation Imaging for the Evaluation of Treatment Response Comparing Three Different Bronchodilator Aerosol Delivery Methods in Patients With COPD: A Pilot Study
Brief Title: Comparison of Bronchodilator Response From Three Different Aerosol Delivery Methods in Patients With COPD Using Hyperpolarized Xe 129 MRI Ventilation Imaging
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Polarean, Inc. (Industry)
Collaborators: Aerogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: POL-Xe-005
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Vibrating Mesh Nebulizer First (Experimental): Participants will receive albuterol delivered via vibrating mesh nebulizer as their first treatment, followed by albuterol delivered via metered dose inhaler and then albuterol delivered via jet nebulizer.
  Interventions: Drug: Albuterol Sulfate, 2.5 Mg/3 mL (0.083%) Inhalation Solution; Device: Vibrating Mesh Nebulizer; Device: Metered Dose Inhaler; Device: Jet Nebulizer
- Jet Nebulizer First (Experimental): Participants will receive albuterol delivered via jet nebulizer as their first treatment, followed by albuterol delivered via vibrating mesh nebulizer and then albuterol delivered via metered dose inhaler.
  Interventions: Drug: Albuterol Sulfate, 2.5 Mg/3 mL (0.083%) Inhalation Solution; Device: Vibrating Mesh Nebulizer; Device: Metered Dose Inhaler; Device: Jet Nebulizer
- Metered Dose Inhaler First (Experimental): Participants will receive albuterol delivered via metered dose inhaler as their first treatment, followed by albuterol delivered via jet nebulizer and then albuterol delivered via vibrating mesh nebulizer.
  Interventions: Drug: Albuterol Sulfate, 2.5 Mg/3 mL (0.083%) Inhalation Solution; Device: Vibrating Mesh Nebulizer; Device: Metered Dose Inhaler; Device: Jet Nebulizer

INTERVENTIONS:
Drug: Albuterol Sulfate, 2.5 Mg/3 mL (0.083%) Inhalation Solution — Aerosolized albuterol
Device: Vibrating Mesh Nebulizer — A vibrating mesh nebulizer will be used to deliver aerosolized albuterol
  Other Names: Solo VMN
Device: Metered Dose Inhaler — A metered dose inhaler will be used to deliver aerosolized albuterol
  Other Names: pMDI-aerosol metered dose inhaler
Device: Jet Nebulizer — A jet nebulizer will be used to deliver aerosolized albuterol
  Other Names: JN nebulizer

SUMMARY:
The goal of this clinical trial is to compare responses to bronchodilator treatment delivered by three different aerosol delivery methods in patients with chronic obstructive pulmonary disease (COPD). The main question it aims to answer is whether there are differences in lung ventilation following treatment with each of the three methods as measured using hyperpolarized Xe 129 with MRI.

Participants will:

Receive a standard dose of albuterol delivered using each of 3 aerosol delivery devices. In total, participants will receive three treatments separated by at least 1 week each.

Following each treatment, participants will have inhale an MRI contrast agent called hyperpolarized Xe 129 and will have images of their lungs taken with an MRI.

Researchers will compare the different lung images taken after each treatment to see if there are differences in the distribution of air in the lungs (known as ventilation).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at enrollment.
2. Participant (or legally acceptable representative) willing and able to provide written informed consent.
3. Able (in the Investigator's opinion) and willing to comply with all study requirements.
4. Documented diagnosis of COPD limited to:

   a. Pulmonary function tests (PFT) value of forced expiratory volume at 1 second/forced vital capacity (FEV₁ / FVC) <70%
5. Receiving standard of care (SOC) background drug therapy as per current guidance for COPD for at least 6 months to screening Visit 1.
6. Participants enrolled as bronchodilator responder:

   a. Increase of ≥12% and ≥200 mL as an absolute value compared with a baseline measure in either forced expiratory volume at 1 second or FVC at screening.
7. Participants enrolled as non-bronchodilator responder:

   a. Increase of ≤12% and ≤200 mL as an absolute value compared with a baseline in either FEV1 or FVC at screening.
8. Stable baseline conditions and no medication changes within 6 weeks of planned imaging visit.
9. Female participants of childbearing potential must be confirmed non-pregnant via serum or dip-stick urine test at baseline (Screening) and prior to each Xe MRI.

Exclusion Criteria:

1. Participant with life expectancy <1-2 years or significant diseases other than COPD.

   A significant disease is defined as a disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the patients' ability to participate in the study.
2. Any condition which, in the opinion of the Investigator, would make it unsafe or unsuitable for the patients to undergo MRI (for example: presence of an implanted or external MRI unsafe device that cannot be removed, body weight exceeding table limitations, inability to lie flat, or severe claustrophobia).
3. Inability to hold breath 10-15 seconds for required imaging or for completion of diffusing capacity of lung for carbon monoxide (DLCO) measurements.
4. Respiratory infection of exacerbation of COPD within the 6 weeks prior to screening.
5. Malignancy for which the patient has undergone resection, radiation, or chemotherapy within the last 5 years. Patients with treated basal cell carcinoma are allowed.
6. Known hypersensitivity to any of the study products.
7. Known or planned pregnancy.
8. Participation in another study which, in the opinion of the Investigator, would interfere with the study compliance, or outcome assessments or would prohibit the collection of the required data points.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percent | measured immediately postdose
  A measure of the percentage of lung area with low ventilation measured using hyperpolarized Xe 129 MRI

SECONDARY OUTCOMES:
Distribution of ventilated space | measured at baseline and immediately postdose
  A measure of distribution of lung ventilation measured using hyperpolarized Xe 129 MRI
Membrane uptake of Xe 129 | measured at baseline and immediately postdose
  A measure of lung membrane air conductance measured using hyperpolarized Xe 129 MRI
Red blood cell Xe 129 transfer | measured at baseline and immediately postdose
  A measure of red blood cell uptake of Xe 129 measured using hyperpolarized Xe 129 MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Mata, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Sheridan Snyder Translational Fontaine Research Unit, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No